CLINICAL TRIAL: NCT04126226
Title: Quality of Life in Patients Treated for Tongue and/or Jaw Neoplasia Before and After Speech Therapy: a Randomized Clinical Trial
Brief Title: Quality of Life in Patients Treated for Tongue and/or Jaw Neoplasia Before and After Speech Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 96487218300005327
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-07

CONDITIONS: Tongue Cancer; Jaw Cancer; Oral Cancer; Intelligibility, Speech
Keywords: Speech therapy; Dysphagia; Speech Intelligibility; Quality of Life
MeSH Terms: conditions — Tongue Neoplasms; Jaw Neoplasms; Mouth Neoplasms; Speech Intelligibility; Communication Disorders; Deglutition Disorders | interventions — Deglutition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental)
  Interventions: Other: Speech-language guidance; Other: Speech therapy exercises for swallowing; Other: Speech therapy exercises for speech
- Control Group (No Intervention)

INTERVENTIONS:
Other: Speech-language guidance — Speech-language guidance for speech enhancement and on food management in terms of consistency, volumes, utensils and temperature, beyond the care for safe and efficient swallowing.
  Arms: Study group
Other: Speech therapy exercises for swallowing — Use of lip exercises and facial muscles, laryngeal elevation maneuver and airway protection technique, 5 repetitions 3 times a day for a month.
  Arms: Study group
Other: Speech therapy exercises for speech — Use of over-articulation technique and glottal firmness exercise, 5 repetitions 3 times a day for a month.
  Arms: Study group

SUMMARY:
This study aims to verify the impact of four speech therapy sessions on the Quality of Life of patients treated for malignant tongue and/or jaw cancer, using as measure specific questionnaires of speech and swallowing.

The hypothesis is that after treatment with exercises and speech therapy guidance, patients will present better indicators on Quality of Life related to speech and swallowing.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 Years
* Tongue and/or Jaw Neoplasm
* Submitted to surgical treatment

Exclusion Criteria:

* Under 18 Years
* Cognitive impairment or deficits in language comprehension
* Previous speech therapy intervention
* Recurrence or active disease
* Death during the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Changes in Quality of Life Scores related to swallowing | 1 month
  To measure the changes in Quality of Life related to swallowing it was used the questionnaire Dysphagia Handicap Index (DHI)
Changes in Quality of Life Scores related to speech | 1 month
  To measure the changes in Quality of Life related to speech it was used the questionnaire Speech Handicap Index (SHI)

SECONDARY OUTCOMES:
Changes in Dysphagia Classification | 1 month
  To measure the changes in Dysphagia classification it was used the Fiberoptic Endoscopic Evaluation of Swallowing, exam that evaluate the functionability of swallow. These exams were presented to three judges (speech therapists) that in agreement classified the degree of dysphagia
Changes in Speech Intelligibility Classification | 1 month
  To measure the changes in Speech Intelligibility it was used speech recordings that were analysed by three judges (speech therapists) that in agreement classified the degree of speech intelligibility

CONTACTS AND LOCATIONS:
Overall Officials: Sady S da Costa, PHD, Study Director — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No